CLINICAL TRIAL: NCT01873547
Title: Different Efficacy Between Rehabilitation Therapy and Umbilical Cord Derived Mesenchymal Stem Cells Transplantation in Patients With Chronic Spinal Cord Injury in China
Brief Title: Different Efficacy Between Rehabilitation Therapy and Stem Cells Transplantation in Patients With SCI in China
Acronym: SCI-III
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: General Hospital of Chinese Armed Police Forces (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013-03-04SCI-III
Record Dates: First submitted 2013-06-04; First posted 2013-06-10 (Estimated); Last update posted 2018-05-25 (Actual); Status verified 2018-05

CONDITIONS: Spinal Cord Injury
Keywords: spinal cord injury; cell transplantation; rehabilitation
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Cell- and Tissue-Based Therapy; Rehabilitation

STUDY DESIGN:
Intervention Model Description: cell therapy or rehabitation treatment
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- rehabilitation (Active Comparator): Patients in the group accept rehabilitation for three weeks in hospital and other eleven months in their home under the guidance of physical therapist.
  Interventions: Other: rehabilitation
- cell therapy (Experimental): Patients in the group accept cell therapy including four times stem cells transplant via intrathecal injection.
  Interventions: Biological: cell therapy
- control (No Intervention): Patients receive no professional treatment in hospital or rehabilitation centre.

INTERVENTIONS:
Biological: cell therapy — Mesenchymal stem cells derived from umbilical cord are transplanted directly into subarachnoid by Lumbar puncture.
  Arms: cell therapy
Other: rehabilitation — Patients only receive rehabilitation of limb function.
  Other Names: physical exercise rehabilitation
  Arms: rehabilitation

SUMMARY:
The morbidity of spinal cord injury (SCI) is increasing year by year significantly in China. The methods to treat SCI patients in sequela stage update are poor. Though traditional rehabilitation therapy is the routine method to treat SCI in sequela stage, aiming to improve the neurological disorders of these patients, such as sensory disturbance, dyskinesia, autologous adjustment of blood pressure, dysfunction of urination, defecation and perspiration , etc. What's a pity, the efficacy of the rehabilitation therapy is unsatisfactory. Rehabilitation Therapy can prevent the process of muscle atrophy and joint stiffness. However, it can not repair the damaged nerve function. Studies show that mesenchymal stem cell transplantation can remarkably improve the neurological function of SCI in animals without any severe side effect.

In this study, 300 patients will be divided into three groups and the investigators will use mesenchymal stem cells derived from umbilical cord to treat 100 SCI patients. They will also follow up 100 patients who only receive rehabilitation and another 100 patients who accept neither stem cell therapy nor rehabilitation. On this basis, the investigators can compare the efficacy of these two treatments.

DETAILED DESCRIPTION:
Patients enrolled in this study need to finish our whole follow-up survey, which is carried out by clinical doctors and epidemiologist.

ELIGIBILITY:
Inclusion Criteria:

1. Patients or their curator must be able to give voluntary consent.
2. Patients have clear history of traumatic injury.
3. 20 years - 65 years of age can be enrolled.
4. Both male and female can be enrolled.
5. The diagnosis of spinal cord injury are confirmed by all of the examinations including MRI, electromyogram and electrophysiology.
6. The time of injury was longer than 1 year.

Exclusion Criteria:

1. Mental disorders
2. Myelitis
3. Women in pregnancy
4. Cancer

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2012-06; Primary Completion 2014-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Assessment of changes in International Standards for Neurological Classification of Spinal Cord Injury according to American Spine Injury Association | Baseline, 6 and 12 months after recruitment
  ASIA is American Spine Injury Association.The ASIA publishes the International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI), which is a neurological exam widely used to document sensory and motor impairments following spinal cord injury (SCI). The ASIA assessment is the gold standard for assessing SCI. The exam is based on neurological responses, touch and pinprick sensations tested in each dermatome, and strength of the muscles that control key motions on both sides of the body. Muscle strength is scored on a scale of 0-5 according to the adjacent table, and sensation is graded on a scale of 0-2: 0 is no sensation, 1 is altered or decreased sensation, and 2 is full sensation. Each side of the body is graded independently. The ISNCSCI exam is used for determining the neurological level of injury. ASIA Impairment Scale for classifying spinal cord injury includes five grades: A, B, C, D and E.

SECONDARY OUTCOMES:
Assessment of changes in score of pain index using Short-form McGill Pain Questionnaire | Baseline,6 and 12 months after recruitment
  The McGill Pain Questionnaire (MPQ) is an international standard scale for description and evaluation of pain.The Short-form McGill Pain Questionnaire (SF-MPQ) is simplified on the basis of MPQ and has high reliability in clinical applications.The main component of the SF-MPQ consists of 15 descriptors (11 sensory; 4 affective) which are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate or 3 = severe. Three pain scores are derived from the sum of the intensity rank values of the words chosen for sensory, affective and total descriptors.
Assessment of changes in score of activity of daily living | Baseline, 6 and 12 months after recruitment
  Bathal Index (BI) is one of the most commonly used methods for measuring the activity of daily living. The BI consists of a 0 - 10 scale measuring discomfort, pain, and fatigue (0 being no problem and 10 being the worst problem) in response to six questions asked of the patient pertaining to the five major symptoms of spinal cord injury: (1)Fatigue; (2)Spinal pain; (3)Arthralgia (joint pain) or swelling; (4)Enthesitis, or inflammation of tendons and ligaments (areas of localized tenderness where connective tissues insert into bone); (5)Morning stiffness duration; (6)Morning stiffness severity.
Assessment of changes in sensory evoked potentials and motor evoked potentials | Baseline,6 and 12 months after recruitment
  A bipolar electrode was placed at 2-3 cm near the distal end of the wrist wrinkle to stimulate the median nerve. An anode was placed near the proximal end. Electrodes for recording were placed at the ipsilateral supraclavicular fossa (Erb') and 1-2 cm above the spinous process of C7 and C4' (for recording of somatosensory evoked potential on the left median nerve) or C3' (for recording of somatosensory evoked potential on the right median nerve). Recordings were made separately on the left and right sides. 200 potentials on each body side were recorded and superimposed. Results of recordings will show whether the latency is apposite or similar with normal.

CONTACTS AND LOCATIONS:
Overall Officials: Yihua An, Ph.D, Study Director — the General Hospital of Chinese People's Armed Police Forces
Locations (1):
- General Hospital of Chinese People's Armed Police Forces, Beijing, Beijing Municipality, China